CLINICAL TRIAL: NCT06439472
Title: Effectiveness of the Suboccipital Inhibition Technique in Individuals With Forward Head Posture: Randomized Controlled Trial
Brief Title: Effectiveness of the Suboccipital Inhibition Technique in Forward Head Posture.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OST1_016
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Individuals With Forward Head Posture
Keywords: Forward head posture; Craniovertebral angle; Suboccipital muscles; Osteopathy.

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Dual (participant, outcome assessor). Participants will be assigned codes, these codes will be randomized via the website https://www.invertexto.com/numeros-aleatorios, and randomly distributed into two groups, a control group and an experimental group, where only the principal investigator and the care provider will have access.
  The outcome assessors will also have no contact with the researcher and the participant during the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suboccipital Inhibition Technique (Experimental): Experimental: Suboccipital Inhibition Technique
  Interventions: Other: Suboccipital Inhibition Technique
- Sham Technique (Placebo Comparator): Placebo Comparator: Sham Technique
  Interventions: Other: Sham Technique

INTERVENTIONS:
Other: Suboccipital Inhibition Technique — The researcher will place their palms under the patient's head and use their fingers to contact the occipital condyles. Next, the researcher will place the 3rd and 4th fingers of each hand in the space between the occiput and the spinous process of C2. The metacarpophalangeal joints are at 90º flexion, with the base of the skull resting on their hands while they apply constant, non-painful pressure in a postero-anterior direction, keeping the 2nd, 3rd and 4th fingers together in extension. Afterwards, the researcher applies a light and gentle traction in a cephalad direction in order to relieve the suboccipital area. Once the suboccipital muscles have relaxed, the researcher gently removes the contact, leaving the participant's head resting on the table.
  This technique is performed for 4 minutes.
  Arms: Suboccipital Inhibition Technique
Other: Sham Technique — The participant is instructed to lie down in the supine position while the mediator assumes a position at the head of the table and places their hands on the participant's shoulders. This technique is performed for 4 minutes.
  Arms: Sham Technique

SUMMARY:
In this randomized controlled experimental trial, it is aimed to verify the effectiveness of applying the suboccipital inhibition technique in altering forward head posture, increasing the craniovertebral angle and decreasing the angle between the chin, the external acoustic meatus and the sternal angle.

DETAILED DESCRIPTION:
Forward head posture (FHP) is defined as misalignment of the head caused by anterior translation of the head in relation to the trunk, The incidence rate of this postural alteration is 66% in individuals between the ages of 20 and 50.

In order to diagnose this alteration, two angles are used: the craniovertebral angle (CVA) and the angle between the chin, the external acoustic meatus and the sternal angle (AMME), with the CVA being the reference angle for diagnosing a FHP. According to the literature, when the CVA is less than 49.9º, there is a FHP.

We decided to use the suboccipital inhibition technique, which according to Eileen DiGiovanna et al (2005), causes a decrease in muscle tension leading to their relaxation. This relaxation, according to Heredia Rizo et al (2012), has significant effects on increasing CVA, which in turn will decrease AMME, resulting in a positive change in FHP.

ELIGIBILITY:
Inclusion Criteria:

* male and female;
* be over 18 years old;
* have a craniovertebral angle of less than 49.9º.

Exclusion Criteria:

* have a craniovertebral angle greater than 49.9º;
* be a 3rd or 4th year osteopathy student;
* be an osteopath.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral angle | Immediately after the intervention.
  To obtain the craniovertebral angle, the SAPO postural assessment software will be used. This angle will be measured in the sagittal plane, with the participant sitting on a chair with their feet shoulder-width apart, resting on the floor, forearms relaxed over their legs, looking at a fixed point positioned on the wall 1 meter in front of their eyes.
  The SAPO software will determine the angle measurement. This procedure will be carried out 3 times in order to minimize the reading error.
Angle between the chin, external acoustic meatus and the sternal angle. | Immediately after the intervention.
  To obtain this angle, the SAPO postural assessment software will be used. This angle will be measured in the sagittal plane, with the participant sitting on a chair with their feet shoulder-width apart, resting on the floor, forearms relaxed over their legs, looking at a fixed point positioned on the wall 1 meter in front of their eyes.
  The SAPO software will determine the angle measurement. This procedure will be carried out 3 times in order to minimize the reading error.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior de Saúde do Porto
Locations (1):
- Escola Superior de Saúde do Porto, Porto, Portugal

REFERENCES:
- [Background] Aggarwal, A., Nair, A., Palekar, TJ e Bhamare, D. (2022). Efeito da técnica de liberação suboccipital na postura anterior da cabeça: um estudo comparativo. Jornal Médico da Universidade Dr. DY Patil , 15 (4), 534-537.
- [Background] Contractor, ES, Shah, S. e Dave, P. (2019). Estudar o efeito imediato da técnica de energia muscular suboccipital no ângulo craniovertebral e no ângulo crânio-horizontal em indivíduos com postura de cabeça anteriorizada. Int J Health Sci Res , 9 (3), 83.
- [Background] Kim, BB, Lee, JH, Jeong, HJ e Cynn, HS (2016). Efeitos da liberação suboccipital com exercício de flexão craniocervical no alinhamento craniocervical e na atividade muscular cervical extrínseca em indivíduos com postura anterior da cabeça. Jornal de Eletromiografia e Cinesiologia , 30 , 31-37.
- [Background] Weber, P., Corrêa, ECR, Milanesi, JM, Soares, JC, & Trevisan, ME (2012). Postura craniocervical: análise cefalométrica e biofotogramétrica. Revista Brasileira de Ciências Orais , 11 (3), 416-421.
- [Background] DiGiovanna, E. L., Schiowitz, S., Dowling, D. J. (2005). Uma abordagem osteopática para diagnóstico e tratamento. Lippincott Williams & Wilkins.